CLINICAL TRIAL: NCT00992940
Title: A Comparison of Patient-controlled Versus Anesthesiologist-controlled Propofol-remifentanil in Awake Craniotomy for Tumor Surgery
Brief Title: Patient-controlled Versus Anesthesiologist-controlled Propofol-remifentanil in Awake Craniotomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds needed to carry on the project were not secured.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0492-A
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Awake Craniotomy for Brain Tumour Surgery
Keywords: awake craniotomy; patient-controlled sedation analgesia; anesthetist-controlled sedation analgesia; remifentanil-propofol; tumour surgery
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-Controlled Sedation/Analgesia (Experimental): Patient controls the amount of sedation and analgesia delivered, according to their own requirements.
  Interventions: Procedure: Patient-Controlled Sedation/Analgesia
- Anesthetist-Controlled Sedation/Analgesia (Active Comparator): Patient sedation and analgesia requirements are delivered by the anesthetist.
  Interventions: Procedure: Anesthetist-Controlled Sedation/Analgesia

INTERVENTIONS:
Procedure: Patient-Controlled Sedation/Analgesia — Patient controls delivery of sedation and analgesia requirements.
  Arms: Patient-Controlled Sedation/Analgesia
Procedure: Anesthetist-Controlled Sedation/Analgesia — All sedation and analgesia requirements are determined and delivered by the attending anesthetist.
  Arms: Anesthetist-Controlled Sedation/Analgesia

SUMMARY:
Awake craniotomy for removal of brain tumour is performed because the tumour may be located close to areas of the brain that control specific functions such as movement or speech. Local anaesthesia (freezing) and sedation are required to make the patient comfortable and free of pain, but also to be able to cooperate for testing of brain function (speaking, moving) in order to preserve these areas while removing the brain tumour. The patient will be administered routine anesthetic drugs (sedatives (propofol) and pain killers (remifentanil)). The amount of sedation and analgesia (pain killer) is individually tailored to each patient as each person has different requirements. The usual way to give these medications is by the anesthesiologist assessing pain level, watching the patient and monitoring blood pressure and heart rate. Another way to give this medication is now available. This is with a special device, known as a patient-controlled analgesia pump (PCA). This device allows the patient to push a button to give pain medicine through an intravenous line and is frequently used for pain treatment after surgery and for other types of procedures. This device may be helpful during awake craniotomy, as it would allow patient-controlled administration of pain medicine and relaxing medicine whenever required. The amount of medication can be increased by more presses of the pump. At all times during the operation, the anesthesiologist will monitor the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients more than 18 years of age
2. ASA I, II or III
3. Scheduled to undergo awake craniotomy for elective supratentorial tumor resection.

Exclusion Criteria:

1. patients with allergy to the drugs being used.
2. patients at risk for pulmonary aspiration eg patients with history of GERD, gastroparesis (eg diabetic) and obesity.
3. patients with BMI 35 or above
4. patients with severe cardiovascular or respiratory diseases (ASA IV or higher).
5. patients who are pregnant.
6. patients with alcohol or substance abuse.
7. patients who could not understand the concept of PCSA.
8. patients who do not understand and are unable to follow instructions for the study due to a language barrier
9. lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To assess the ability of patient-controlled sedation/analgesia remifentanil-propofol to maintain appropriate levels of sedation and analgesia in commensuration with the needs of the surgery at different stages. | 2 hours, 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Manninen, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada